CLINICAL TRIAL: NCT01413646
Title: Effects of Walnuts on Endothelial Function in Overweight Adults With at Least One Factor of Metabolic Syndrome: A Randomized, Controlled, Cross-Over Trial
Brief Title: Effects of Walnuts on Endothelial Function in Overweight Adults With at Least One Factor of Metabolic Syndrome
Acronym: Walnut2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, David Katz, MD, PRINCIPAL INVESTIGATOR, Griffin Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2009-15
Record Dates: First submitted 2011-07-11; First posted 2011-08-10 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Metabolic Syndrome
Keywords: obesity; walnuts; endothelial function
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut Supplementation (Experimental): Eight weeks with walnut supplementation to an ad lib diet
  Interventions: Dietary Supplement: Walnut Supplementation
- 2 (Placebo Comparator): Eight weeks ad lib diet without walnut supplementation
  Interventions: Dietary Supplement: No walnut supplementation

INTERVENTIONS:
Dietary Supplement: Walnut Supplementation — Eight weeks of walnut supplementation
  Arms: Walnut Supplementation
Dietary Supplement: No walnut supplementation — Eight weeks without walnut supplementation
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of walnut consumption on endothelial function and lipid markers in overweight patients with at least one factor of metabolic syndrome as compared to the control group.

DETAILED DESCRIPTION:
The prevalence of obesity in both adults and children in the United States has increased significantly over the past 50 years. More than 66% of adults in the US are now overweight or obese and at least 17% of children in the population at large are now considered overweight.Obesity may be a factor predisposing patients to a myriad of comorbidities that increase the associated mortality rate.Several large prospective trials have documented that obesity is an independent risk factor for mortality from cardiovascular disease (CVD). Considering the major metabolic and biochemical changes that occur in obesity, such as atherogenic dyslipidemia, insulin resistance and hyperinsulinemia, endothelial dysfunction, and chronic inflammatory and prothrombotic states, obesity plays a role in the pathogenesis of systemic atherosclerosis and its clinical complications.

Walnuts are rich in alpha-linolenic acid, an essential omega-3 fatty acid, L-arginine and antioxidants. Polyunsaturated fatty acids and antioxidants have anti-oxidative effects and are thought to help preserve the endothelium's capacity to generate nitric oxide (NO), which acts to promote vasodilation, stabilize platelets, and promote the anti-inflammatory abilities of the endothelium. Evidence of this anticipated effect would have implications for strategies to prevent or retard type 2 diabetes mellitus and cardiovascular disease. Endothelial function testing using high frequency ultrasound imaging of the brachial artery to assess endothelium-dependent flow-mediated dilatation (FMD) offers a non-invasive, uniquely valuable means of assessing aggregated influences on cardiac risk by gauging a physiologic response of the vascular endothelium. Proposed, therefore, is a randomized, controlled, cross-over clinical trial, to assess the effects of walnuts on endothelial function in overweight adults with elevated waist circumference and at least one risk factor of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age 25-75 years
* Non-smoker
* Overweight (BMI ≥ 25) with central adiposity as indicated by waist circumference (102 cm. in men / 88 cm. in women)
* Meet one risk factor of the metabolic syndrome.

  * blood pressure > 130/85 or taking antihypertensive medication

    * fasting plasma glucose (FPG) >100 mg/dL (6.1 mmol/L)
    * fasting serum triglycerides level (TG) > 150 mg/dL (1.69 mmol/L)
    * fasting high-density lipoprotein (HDL) cholesterol < 40 mg/dL (1.04 mmol/L)in men, and < 50 mg/dL (1.29 mmol/L) in women.

Exclusion Criteria:

* Anticipated inability to complete or comply with study protocol
* Use of lipid-lowering or antihypertensive medications or aspirin unless stable on medication for at least 3 months and willing to refrain from taking medication for 12 hours prior to EF scanning
* Preexisting cardiovascular disease (including symptomatic coronary artery disease (CAD), myocardial infarction, angina pectoris, anginal equivalent, peripheral vascular disease, congestive heart failure, carotid stenosis)
* Severe hypertension (systolic blood pressure >180mmHg or diastolic blood pressure >105mmHg), even if well-controlled by medication.
* Diagnosed diabetes mellitus
* Regular use of multivitamins, Vitamin C, Vitamin E, fish oil, flax seed oil, omega-3 fatty acids, CoQ10, fiber supplements, garlic pills, arginine, red yeast rice, and any kind of antioxidant and unwillingness to discontinue supplementation for at least 4 weeks prior to study initiation and for study duration
* Allergic to walnuts or any other nuts
* Diagnosed eating disorder
* On any specific diet, weight control diet, vegan diet
* Any rheumatologic disease requiring regular use of NSAIDs or alternative medications
* Regular use of fiber supplements
* Regular use of vasoactive medication (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators), and anticoagulant drugs (including Coumadin, plavix )
* Diagnosed sleep apnea
* Substance abuse (chronic alcoholism, other chemical dependency)
* Any unstable medical condition that would limit the ability of a subject to participate fully in the trial (e.g., cancer, AIDS, tuberculosis, psychotic disorder)
* Current or impending pregnancy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 8 weeks
  Brachial artery flow mediated dilation (FMD)

SECONDARY OUTCOMES:
Weight | 8 weeks
Waist circumference | 8 weeks
Fasting lipid panel | 8 weeks
  Total cholesterol, low density lipoprotein cholesterol, high density lipoprotein cholesterol, triglyceride level, cholesterol / high density lipoprotein cholesterol ratio
Fasting blood glucose | 8 weeks
Fasting insulin | 8 weeks
Blood pressure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David L. Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

REFERENCES:
- [Derived] Katz DL, Davidhi A, Ma Y, Kavak Y, Bifulco L, Njike VY. Effects of walnuts on endothelial function in overweight adults with visceral obesity: a randomized, controlled, crossover trial. J Am Coll Nutr. 2012 Dec;31(6):415-23. doi: 10.1080/07315724.2012.10720468. PMID 23756586